CLINICAL TRIAL: NCT05551377
Title: The Heads-Up Trial: Sleeping in a Head-Up Tilt Position to Alleviate Orthostatic Hypotension, Supine Hypertension and Nocturia in Parkinson's Disease
Brief Title: Head-up Tilt Sleeping to Alleviate Orthostatic Hypotension, Supine Hypertension and Nocturia in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL.80610.091.22; MJFF-020200 (Other Grant/Funding Number: Michael J Fox Foundation for Parkinson's Research)
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: Parkinson's disease; Orthostatic hypotension; Supine hypertension; Autonomic dysfunction
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Hypotension, Orthostatic; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: Participants are divided into two groups, the intervention and control (delayed intervention) group.
Who Masked: Participant, Investigator
Masking Description: Both the investigator and the participants are blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): At T0, in-clinic inclusion, we will record basic characteristics and several questionnaires, we will also perform a short tilt-table-test and standing blood pressure (BP) test. Intake is followed by one week of horizontal sleeping for baseline home-based BP measurements. Participants in the intervention group will then sleep in a head-up tilt position for two weeks each in angles 6°, 12° and 18°. At the second and final in-clinic meeting, at T1, measurements done at T0 will be repeated, complemented with an assessment of barriers and facilitators of HUTS. During HUTS daily BP measurements will be done, and data will be collected on orthostatic tolerance, nighttime urine production, subjective comfort of HUTS, falls.
  Interventions: Other: Head-up tilt sleeping
- Delayed intervention group (Other): Follows the same structure as the intervention group, but starts with a HUTS placebo angle of 1° for two weeks, followed by two intervention angles of 6° and 12° for two weeks each. The 1°-angle serves as the control intervention.
  Interventions: Other: Head-up tilt sleeping

INTERVENTIONS:
Other: Head-up tilt sleeping — Whole-body head-up tilt sleeping (HUTS) will be carried out in three different angles, each for the duration of two weeks. Prior to the first angle the participant will sleep in a horizontal position for 1 week. The different angles will be installed using a wedge between the mattress and bed frame.

SUMMARY:
Autonomic dysfunction is common and often underrecognized in Parkinson's disease (PD). Orthostatic hypotension (OH) affects up to a third of PD patients and often coincides with supine hypertension. This co-occurrence complicates pharmacological treatment as treatment of one can negatively affect the other. Head-up tilt sleeping (HUTS) could improve both. This phase II randomized controlled trial (RCT) aims to investigate the efficacy and tolerability of this understudied intervention, leading to optimal implementation strategies.

DETAILED DESCRIPTION:
Autonomic dysfunction is common and often underrecognized in Parkinson's disease (PD). Orthostatic hypotension (OH) affects up to a third of PD patients and about half of them also exhibit supine hypertension. In current clinical practice both are undertreated. The common co-occurrence of OH and supine hypertension complicates pharmacological treatment as improvement of one can be accomplished only at the expense of the other. Head-up tilt sleeping (HUTS) is the only intervention known that could improve both. The concept of HUTS is based on several small-scale observational studies and expert opinion. Although HUTS has been proposed as an effective and even first choice non-pharmacological treatment for OH for over three decades, it is often not advised to patients because of lack of evidence on its effectiveness and on how to implement it. The Heads-Up trial is a multicenter home-based double-blind phase II RCT. The study aims to investigate the efficacy and tolerability of HUTS, leading to optimal implementation strategies of HUTS to treat orthostatic hypotension and supine hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Orthostatic hypotension defined as a systolic BP decrease of ≥20 mmHg, or a diastolic decrease of ≥10 mmHg, within 3 min after changing from a supine to standing position OR mean standing BP of ≤75 mmHg (marker for symptomatic orthostatic hypotension). In patients with supine hypertension, a decrease in systolic BP of ≥ 30 mmHg is required;
* Orthostatic intolerance: direct complaints (dizziness, blurry vision, etc.) and/or indirect signs (falls or freezing episodes that relate to postural challenge);
* Supine hypertension defined as a systolic BP of ≥140 mmHg, and/or diastolic of ≥90 mmHg, after 5 min of supine rest;
* Idiopathic PD or parkinsonism (multiple system atrophy, progressive supranuclear palsy, corticobasal degeneration, vascular parkinsonism and Lewy body dementia);
* Ability to walk (with or without a walking aid), as subjectively determined by the researcher;
* Stable medication regimens for orthostatic hypotension and supine hypertension during the trial;

Exclusion Criteria:

* Inability to follow instructions and complete questionnaires, as assessed by the researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Average overnight supine blood pressure | Measured four times: in week 1, 3, 5 and 7
  Average overnight supine blood pressure (mmHg) from the 24h ambulatory blood pressure measurement (ABPM)

SECONDARY OUTCOMES:
Daily supine blood pressure | Daily in week 1 up to and including week 7
  Supine blood pressure (mmHg) measured every morning directly after awakening before getting out of bed
Orthostatic blood pressure | Measured six times: in-clinic (T0; pre-intervention), in week 1, 3, 5 and 7, and in-clinic on the day after week 7 ends (T1; post-intervention)
  Standing orthostatic blood pressure test (mmHg). Measured in clinic and home-based guided by a researcher via video call.
24h ABPM parameters | In week 1, 3, 5 and 7
  24h ABPM parameters blood pressure variability (mmHg), nocturnal blood pressure dipping (mmHg) and average daytime blood pressure (mmHg). Each of these measures will be derived from the 24 hour blood pressure measurements, and reported separately.
Orthostatic tolerance | Week 1, 3, 5 and 7
  Self-reported burden of symptoms of orthostatic hypotension (Orthostatic hypotension questionnaire (OHQ)). The score ranges from 0 to 100, with a higher number meaning worse symptoms of orthostatic hypotension.
Nocturia | Week 1, 3, 5 and 7
  Self-reported frequency of daytime and night time urination and impact on quality of life (International Consultation on Incontinence Questionnaire Nocturia Module (ICIQ-N))
Subjective comfort of HUTS (head up tilted sleeping) | Week 1, 3, 5 and 7
  Self-reported tolerability of the head up tilted sleeping at different angles including questions about sleep duration, sleep quality and comfort, and feeling rested in the morning.
Falls | Week 1, 3, 5 and 7
  Self-reported falls and in case of a fall additional questions about the time and circumstances
Overnight change in body weight | Daily in week 1 up to and including week 7
  Weight (kg) difference between the evening and the morning, both measured after micturition
Nighttime urine production | Week 1, 3, 5 and 7
  Urine volume measured in a urinal (ml)
Barriers and facilitators of the intervention | Immediately post-intervention (day after week 7, T1)
  Structured interview

OTHER OUTCOMES:
Timed up and go test (TUG) | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Measurement of the time that the participant takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees
Symptoms of Parkinson's disease | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Movement disorders society unified disease rating scale (MDS-UPDRS). Scores range from 0 to 199, with a higher score indicating a more severe impairment related to Parkinson's disease.
Quality of sleep | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Pittsburgh Sleep Quality Index (PSQI). Score ranges from 0 to 21, with 21 indicating a worse sleep quality.
Fear of falling | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Falls Efficacy Scale (FES). Scores ranges from 16 to 67, with a higher score meaning a worse fear of falling.
Subjective level of physical activity | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Longitudinal Aging Study Amsterdam (LASA) Physical Activity Questionnaire (LAPAQ). Score corresponds to time spend doing physical activities. A higher score indicates a more active last two weeks.
Cardiovascular autonomic symptoms | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Selected cardiovascular questions from the Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT). Scored 0 to 9, a worse score means more symptoms of orthostatic hypotension.
Experienced quality of life | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Quality of life questionnaire: the Parkinson's disease questionnaire (PDQ-39). Scores range from 0 to 100, with a higher score indicating a worse quality of life.
Experienced anxiety and depression | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Quality of life questionnaire: the hospital anxiety and depression scale (HADS). Scores range from 0 to 21 for depression and anxiety, a score between 0-7 means no anxiety or depression, 8-14 possibility of an anxiety or depressive disorder and 15-21 likely a depressive or anxiety disorder.
Mental health | Pre-intervention (day before week 1, T0) and post-intervention (day after week 7,T1)
  Quality of life questionnaire: the Mental Health Continuum-Short Form (MHC-SF). Scores range from 0 to 70, with a higher score meaning a better emotional wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Roland D Thijs, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Relevant and anonymized research data will be shared in the validated research database DANS Easy (Data Archiving and Networked Services). It will also be shared with the funding foundation (MJFF).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Study protocol and statistical analysis plan are shared with the funding foundation prior to the onset of the study. After completion of the measurements and analysis we will share the clinical study report with the funding foundation and place relevant and anonymized data on the DANS Easy database.
Access Criteria: Access to the data is restricted, meaning that researchers who are interested in re-use of the data are asked to contact the central contact person for permission. Approval is given after a signed agreement.

REFERENCES:
- [Derived] van der Stam AH, de Vries NM, Shmuely S, Smeenk D, Rutten JH, van Rossum IA, de Bot ST, Claassen JA, Bloem BR, Thijs RD. Study protocol for the Heads-Up trial: a phase II randomized controlled trial investigating head-up tilt sleeping to alleviate orthostatic intolerance in Parkinson's Disease and parkinsonism. BMC Neurol. 2024 Jan 2;24(1):4. doi: 10.1186/s12883-023-03506-x. PMID 38166676